CLINICAL TRIAL: NCT05246540
Title: Evaluation of PET/CT of Cephalic Arteries for the Diagnosis of Giant Cell Arteritis
Acronym: Cervico-TEP et
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: ALBERINI CHU 2020
Record Dates: First submitted 2022-02-09; First posted 2022-02-18 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Giant Cell Arteritis
MeSH Terms: conditions — Giant Cell Arteritis | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Data collection

SUMMARY:
Giant cell arteritis (GCA) is the most common vasculitis in adults. The diagnosis of GCA is evoked by the association of clinical signs and biological anomalies (inflammatory syndrome) in patients over 50 years of age. On the other hand, starting a treatment implies being certain of the diagnosis which requires performing a temporal artery biopsy under local anesthesia. This examination is therefore an invasive procedure for patients whose sensitivity is not optimal. This is why imaging techniques (echo-Doppler or MRI of the temporal arteries) have been developed to look for signs of vasculitis without the need to perform a biopsy. However, these examinations lack sensitivity (=falsely concluding the absence of GCA) and specificity (=falsely concluding the presence of GCA). Recently, advances in imaging, and in particular positron emission tomography (PET), have made it possible to visualize the cephalic arteries, including the temporal artery.

The aim of this study is therefore to evaluate the sensitivity and specificity of PET of the cephalic arteries for the diagnosis of GCA and to compare them with those of echo-Doppler and MRI of the temporal arteries.

ELIGIBILITY:
Inclusion Criteria:

* Any patient for which the diagnosis of GCA is suspected and who underwent a cervical PET/CT

Exclusion Criteria:

* previously diagnosed GCA, glycemia > 7 mmol/L, PET CT performed more than 72 h after introduction of glucocorticoids, age < 50 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: outpatient
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Sensitivity / specificity of cervical PET/CT for the diagnosis of GCA | 6 months
  diagnosis retained by the clinician without question after 6 months of follow-up and treatment for at least 6 consecutive months

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France

REFERENCES:
- [Result] Thibault T, Durand-Bailloud B, Soudry-Faure A, Greigert H, Drouet C, Devilliers H, Ramon A, Bejot Y, Martin L, Creuzot-Garcher C, Falvo N, Audia S, Cochet A, Bonnotte B, Alberini JL, Samson M. PET/CT of cranial arteries for a sensitive diagnosis of giant cell arteritis. Rheumatology (Oxford). 2023 Apr 3;62(4):1568-1575. doi: 10.1093/rheumatology/keac430. PMID 35866984